CLINICAL TRIAL: NCT02393716
Title: Endurant Evo US Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study terminated enrollment due to device failures prior to enrollment completion.
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10173341DOC
Record Dates: First submitted 2015-03-06; First posted 2015-03-19 (Estimated); Results first posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Abdominal Aortic Aneurysm; AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Endovascular repair (Other): Endurant Evo AAA Stent Graft System
  Interventions: Device: Endurant Evo AAA Stent Graft System; Procedure: Endovascular aneurysm repair (EVAR)

INTERVENTIONS:
Device: Endurant Evo AAA Stent Graft System
Procedure: Endovascular aneurysm repair (EVAR)

SUMMARY:
The purpose of this study is to demonstrate that the Endurant Evo Abdominal Aortic Aneurysm (AAA) stent graft system is safe and effective for endovascular treatment of infrarenal abdominal aortic or aortoiliac aneurysms.

DETAILED DESCRIPTION:
The clinical evidence collected as part of this trial will be used in conjunction with data collected during the concurrently enrolling Endurant Evo International Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years old
2. Subject understands and voluntarily has signed and dated the Informed Consent approved by the Sponsor and by the Ethics Committee/Institutional Review Board
3. Subject is able and willing to comply with the protocol and to adhere to the follow-up requirements
4. Subject is a suitable candidate for elective surgical repair of AAA as evaluated by American Society of Anesthesiologists (ASA) Physical Status Classification System I, II, or III
5. Subject has an infrarenal abdominal aortic or aortoiliac aneurysm characterized by one or more of the following:

   * Aneurysm is >5 cm in diameter (diameter measured is perpendicular to the line of flow)
   * Aneurysm is 4 - 5 cm in diameter and has increased in size ≥0.5 cm within the previous 6 months
6. Subject meets all the following anatomical criteria as demonstrated on contrast-enhanced computed tomography (CTA) or magnetic resonance angiography (MRA) imaging:

   * Proximal neck length of ≥ 10 mm with ≤ 60° infrarenal and ≤ 45° suprarenal neck angulation or Proximal neck length of ≥ 15 mm with ≤ 75° infrarenal and ≤ 60° suprarenal neck angulation
   * Subject has vascular dimensions, e.g., aortic and iliac diameters, lengths from renal arteries to iliac bifurcation and hypogastric arteries, in the range of sizes available for the Endurant Evo AAA stent graft system (measured intima to intima) and within the sizing recommendations (refer to Endurant Evo AAA stent graft system Instructions for Use (IFU))
   * Subject has a proximal aortic neck diameter ≥ 18 mm and ≤ 32 mm
   * The distal fixation center of the iliac arteries must have a diameter ≥ 7 mm and ≤ 25 mm bilaterally for the bifurcation and unilaterally for the Aorto-uni-iliac stent graft (AUI)
   * Subject has documented imaging evidence of at least one patent iliac and one femoral artery, or can tolerate a vascular conduit that allows introduction of the Endurant Evo AAA stent graft system
   * Subject has distal non-aneurysmal iliac (cylindrical) fixation length ≥20 mm bilateral for the bifurcation and unilaterally for the AUI

Exclusion Criteria:

1. Subject has a life expectancy ≤1 year
2. Subject is participating in another investigational drug or device study which would interfere with the endpoints and follow-ups of this study
3. Subject is pregnant
4. Subject has an aneurysm that is:

   * Suprarenal/pararenal/juxtarenal
   * Isolated ilio-femoral
   * Mycotic
   * Inflammatory
   * Pseudoaneurysm
   * Dissecting
   * Ruptured
   * Leaking but not ruptured
5. Subject requires emergent aneurysm treatment
6. Subject has a known, untreated thoracic aneurysm >4.5 cm in diameter at the time of screening
7. Subject has been previously treated for an abdominal aortic aneurysm
8. Subject has a history of bleeding diathesis or coagulopathy
9. Subject has had or plans to have an unrelated major surgical or interventional procedure within 1 month before or after implantation of the Endurant Evo AAA stent graft
10. Subject has had a myocardial infarction (MI) or cerebral vascular accident (CVA) within 3 months prior to implantation of the Endurant Evo AAA stent graft
11. Subject has a conical neck defined as a >4 mm distal increase from the lowest renal artery over a 10 mm length
12. Subject has a known allergy or intolerance to the device materials
13. Subject has a known hypersensitivity or contraindication to anticoagulants, antiplatelets, or contrast media, which is not amenable to pre-treatment
14. Subject has significant aortic thrombus and/or calcification at either the proximal or distal attachment centers that would compromise fixation and seal of the device at the discretion of the investigator
15. Subject has ectatic iliac arteries requiring bilateral exclusion of hypogastric blood flow
16. Subject whose arterial access site is not anticipated to accommodate the diameter of the Endurant Evo AAA stent graft delivery system (13F-17F) due to vessel size, calcification, or tortuosity
17. Subject is morbidly obese or has other documented clinical conditions that severely inhibit radiographic visualization of the aorta at the discretion of the investigator
18. Subject has active infection at the time of the index procedure documented by e.g. pain, fever, drainage, positive culture and/or leukocytosis considered to be clinically significant per investigator discretion
19. Subject has congenital degenerative collagen disease, e.g., Marfan's Syndrome
20. Subject has a creatinine level > 2.00 mg/dl (or >176.8 μmol/L)
21. Subject is on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Upchurch, MD, Principal Investigator — University of Florida
Locations (14):
- United States (14):
  - Kaiser Permanente Zion Medical Center, San Diego, California
  - Stanford Hospital & Clinics, Stanford, California
  - Medstar Heart & Vascular Institute, Washington D.C., District of Columbia
  - Maine Medical Center, Portland, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health Sysem, Ann Arbor, Michigan
  - Long Island Jewish Northshore University Hospital, New Hyde Park, New York
  - The Christ Hospital, Cincinnati, Ohio
  - UPMC Pinnacle Harrisburg Campus, Harrisburg, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - University of Virginia, Charlottesville, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Aurora St. Lukes Medial Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Global enrollment was stopped at 139 out of 140 planned. Enrollment start date: 20 April 2015
Groups:
- Endovascular Repair: Endurant Evo AAA Stent Graft System
  Endurant Evo AAA Stent Graft System
  Endovascular aneurysm repair (EVAR)
Period: Overall Study
Arm/Group | Endovascular Repair
Started | 139
Completed | 78
Not Completed | 61
Not completed — Death | 29
Not completed — Withdrawal by Subject | 8
Not completed — Device Explanted | 8
Not completed — Missed visit | 16

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 124
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 70
  Europe | 69

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Experiencing a Major Adverse Event (MAE) Within 30 Days Post-implantation.
Description: The percentage of subjects experiencing a Major Adverse Event (MAE) within 30 days post-implantation.
  MAEs include the occurrence of any of the following events:
  * All-cause mortality
  * Bowel ischemia
  * Myocardial infarction
  * Paraplegia
  * Procedural blood loss ≥1000 cc
  * Renal failure
  * Respiratory failure
  * Stroke
Time Frame: 30-days
Population: Globally, 4 out 139 Subjects experienced a MAE within 30 days (2.9%).
Measure: Count of Participants; unit: Participants
Groups:
- Endovascular Repair: Endurant Evo AAA Stent Graft System
  Endovascular aneurysm repair (EVAR)
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 139
Participants | 4
Statistical Analysis 1: Comparison: Endovascular Repair; The primary safety endpoint was tested against a predetermined safety Performance Goal (PG) using the following statistical hypotheses: H0: p ≥ 20% vs. H1: p < 20% where p is the proportion of subjects experiencing a MAE within 30 days of the index procedure in the target population of subjects treated with the Endurant Evo AAA Stent graft system and 20% is the safety PG; Test type: Other — Single arm study with a hypothesis test comparing to performance goal; p < 0.001, Based on exact binomial distribution; Percentage = 2.9, 97.5% CI 1-sided [upper limit 7.2]

2. Primary Outcome: The Percentage of Subjects With Both Technical Success at the Time of Index Procedure and Treatment Success at 12-months Post-implantation.
Description: Successful aneurysm treatment was achieved based on the following criteria:
  Technical success at the index procedure (as assessed intra-operatively), defined as successful delivery and deployment of the Endurant Evo AAA Stent graft system in the planned location and with no unintentional coverage of both internal iliac arteries or any visceral aortic branches and with successful removal of the delivery system AND
  Treatment success consisting of freedom from:
  * AAA diameter increase, defined as > 5 mm increase in maximum diameter as measured on computed tomography (CT) scan or magnetic resonance angiography/magnetic resonance imaging (MRA/MRI) at 12-month follow-up as compared to 1-month imaging
  * Types I and III endoleaks at 12-month follow-up including those requiring intervention through 12 months
  * Aneurysm rupture within 365 days
  * Conversion to surgery within 365 days
  * Stent graft migration resulting in a serious adverse event or requiring seco
Time Frame: 12-months
Population: While the full 139 subjects were evaluable for Technical Success at index procedure, 118 subjects were evaluable for treatment success at 12 month follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 139
Participants
  Primary Effectiveness (Technical Success) | 139
  Primary effectiveness (Technical Success and treatment Success): number analyzed (Participants) | 118
  Primary effectiveness (Technical Success and treatment Success) | 113
Statistical Analysis 1: Comparison: Endovascular Repair; The primary effectiveness endpoint was tested against a predetermined effectiveness PG using following statistical hypotheses: H0: q ≤ 80% vs. H1: q > 80% where q is the proportion of subjects who have a successful aneurysm treatment in the target population of subjects treated with the Endurant Evo AAA Stent graft system and 80% is the effectiveness PG; Test type: Other — Single-arm study with a hypothesis test comparing to performance goal; p < 0.001, Based on exact binomial distribution; Percentage = 95.8, 97.5% CI 1-sided [lower limit 90.4]

3. Secondary Outcome: All-cause Mortality
Description: All-cause mortality (ACM) within 30, 183, 365 days
Time Frame: within 30, 183, and 365 days
Population: At 0-365 days, 138 subjects were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 139
Participants
  All-Cause Mortality 0-30 Days | 1
  All-Cause Mortality 0-183 Days | 4
  All-Cause Mortality 0-365 Days: number analyzed (Participants) | 138
  All-Cause Mortality 0-365 Days | 8

4. Secondary Outcome: Aneurysm-related Mortality (ARM)
Description: Aneurysm-related mortality (ARM) within 30, 183, and 365 days
Time Frame: within 30, 183, and 365 days
Population: In 0-365 days, 133 subjects were evaluable for Aneurysm related mortality
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 139
Participants
  Aneurysm-related mortality (ARM) 0-30 days | 1
  Aneurysm-related mortality (ARM) 0-183 days | 1
  Aneurysm-related mortality (ARM) 0-365 days: number analyzed (Participants) | 133
  Aneurysm-related mortality (ARM) 0-365 days | 1

5. Secondary Outcome: Secondary Procedures to Correct Type I and III Endoleaks
Description: Any reintervention procedure (surgical or endovascular) following the completion of the operative initial implantation procedure that is used to correct a Type I and III endoleaks within 183 and 365 days. Type I endoleak was defined as a leak resulting from an incomplete seal of the endograft proximally or distally and a Type III endoleak was defined as a leak resulting from a defect of fabric or between the segments of the modular graft (junctional endoleak.
Time Frame: within 183, and 365 days
Population: In 0-183 days, 138 subjects were evaluable In 0-365 days, 132 subjects were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 138
Participants
  0-183 days | 0
  0-365 days: number analyzed (Participants) | 132
  0-365 days | 1

6. Secondary Outcome: Secondary Procedures
Description: Secondary procedures within 183 and 365 days
Time Frame: within 183, and 365 days
Population: In 0-183 days, 138 subjects were evaluable In 0-365 days, 134 subjects were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 138
Participants
  0-183 days | 2
  0-365 days: number analyzed (Participants) | 134
  0-365 days | 6

7. Secondary Outcome: Serious Adverse Events
Description: Serious adverse events within 30, 183 and 365 days.
Time Frame: within 30, 183, and 365 days
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 139
Participants
  0-30 days | 25
  0-183 days | 48
  0-365 days | 60

8. Secondary Outcome: Conversion to Open Surgery
Description: Conversion to open surgery within 183, and 365 days
Time Frame: within 183, and 365 days
Population: In 0-183 days, 138 subjects were evaluable In 0-365 days, 133 were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 138
Participants
  0-183 days | 1
  0-365 days: number analyzed (Participants) | 133
  0-365 days | 2

9. Secondary Outcome: Aneurysm Rupture
Description: Aneurysm rupture within 183 and 365 days
Time Frame: within 183 and 365 days
Population: In 0-183 days, 138 subjects were evaluable In 0-365 days, 132 subjects were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 138
Participants
  0-183 days | 0
  0-365 days: number analyzed (Participants) | 132
  0-365 days | 0

10. Secondary Outcome: Major Adverse Events
Description: Major adverse events within 183 and 365 days
Time Frame: within 183 and 365 days
Population: In 0-183 days, 139 subjects were evaluable In 0-365 days, 138 subjects were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 139
Participants
  0-183 days | 10
  0-365 days: number analyzed (Participants) | 138
  0-365 days | 16

11. Secondary Outcome: Stent Graft Migration
Description: Stent graft movement of either the main body or iliac limb distally or proximally at 6- and 12-month follow-up visits (as compared to 1-month imaging). Main body stent graft migration is defined as evidence of movement of the main body stent graft relative to fixed anatomic landmarks, which is not due to remodeling of the subject's vasculature. Migration is observed when the stent graft completely covers a renal artery or movement is > 10 mm either distally or proximally. Stent graft limb/extension migration is defined as evidence of a movement of the stent graft limbs/extensions relative to fixed anatomic landmarks, which is not due to remodeling of the subject's vasculature that is > 10 mm or coverage of the internal iliac artery.
Time Frame: At 6- and 12-month follow-up visits (as compared to 1-month imaging)
Population: At 6-months, 124 subjects were evaluable At 12-months, 121 subjects were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 124
Participants
  6-months | 1
  12-months: number analyzed (Participants) | 121
  12-months | 2

12. Secondary Outcome: Aneurysm Expansion >5 mm
Description: Aneurysm expansion >5 mm at 6- and 12-month follow-up visits (as compared to 1-month imaging)
Time Frame: at 6- and 12-month follow-up visits (as compared to 1-month imaging)
Population: At 6-months, 130 subjects were evaluable. At 12-months, 123 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 130
Participants
  6-months | 2
  12-months: number analyzed (Participants) | 123
  12-months | 2

13. Secondary Outcome: All Endoleaks Based on Imaging Findings
Description: All endoleaks based on imaging findings at 1-month, 6-month and 12-month. An endoleak is defined by the presence of contrast-enhanced blood outside the lumen of the endoluminal graft but within the aneurysm sac as seen on computed tomography (CT), angiography, ultrasound, or other appropriate imaging modality.
Time Frame: at 1-, 6-, and 12-month follow-up visits
Population: At 1-month 134, subjects were evaluable. At 6-months, 124 subjects were evaluable. 12-months 117 subjects were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 134
Participants
  1-month. Participants with any type of endoleak | 45
  6-months. Participants with any type of endoleak: number analyzed (Participants) | 124
  6-months. Participants with any type of endoleak | 29
  12-months. Participants with any type of endoleak: number analyzed (Participants) | 117
  12-months. Participants with any type of endoleak | 29

14. Secondary Outcome: Stent Graft Occlusions Based on Imaging Findings
Description: Stent graft occlusions based on imaging findings through 1-, 6- and 12 months. Stent graft occlusion is defined as a 100% blockage of the lumen diameter of any implanted stent graft component(s) as evidenced by CT, angiography, ultrasound, or other appropriate imaging modality, and/or operative or pathological analysis.
Time Frame: Through 1-, 6- and 12 months
Population: Through 1-month, 136 subjects were evaluable. Through 6-months, 124 subjects were evaluable. Through 12-months, 120 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 136
Participants
  1-month | 0
  6-months: number analyzed (Participants) | 124
  6-months | 1
  12-months: number analyzed (Participants) | 120
  12-months | 1

15. Secondary Outcome: Device Deficiencies Based on Imaging Findings
Description: Device deficiencies based on imaging findings through 6- and 12 months. A device deficiency was defined according Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance (ref. ISO 14155:2011 3.15).
Time Frame: Through 6- and 12 months
Population: Through 6-months, 125 subjects were evaluable. Through 12-months, 126 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 126
Participants
  6-months. Any device deficiency.: number analyzed (Participants) | 125
  6-months. Any device deficiency. | 27
  12-months. Any device deficiency. | 41

ADVERSE EVENTS:
Time Frame: 60-month
Arm/Group | Endovascular Repair
All-Cause Mortality (participants affected / at risk) | 29/139
Serious Adverse Events (participants affected / at risk) | 105/139
Other Adverse Events (participants affected / at risk) | 38/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Repair (N=139)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Heparin induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 7 (7)
ANGINA PECTORIS (Cardiac disorders) | 3 (3)
ANGINA UNSTABLE (Cardiac disorders) | 3 (4)
AORTIC VALVE STENOSIS (Cardiac disorders) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 7 (9)
BRADYCARDIA (Cardiac disorders) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 3 (3)
CARDIAC FAILURE (Cardiac disorders) | 2 (2)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 2 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 5 (9)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 1 (1)
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1)
INTESTINAL POLYP (Gastrointestinal disorders) | 1 (1)
LOCALISED INTRAABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 3 (3)
CHEST PAIN (General disorders) | 2 (2)
DEATH (General disorders) | 3 (3)
DEVICE DAMAGE (General disorders) | 1 (1)
DEVICE DISLOCATION (General disorders) | 1 (1)
IMPAIRED HEALING (General disorders) | 1 (1)
MALAISE (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
STENT-GRAFT ENDOLEAK (General disorders) | 16 (18)
THROMBOSIS IN DEVICE (General disorders) | 3 (5)
CHOLECYSTITIS (Hepatobiliary disorders) | 3 (3)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 (2)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 (1)
BACTERIAL INFECTION (Infections and infestations) | 2 (2)
BACTERIAL SEPSIS (Infections and infestations) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
GROIN INFECTION (Infections and infestations) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
INFECTIVE ANEURYSM (Infections and infestations) | 1 (1)
INFLUENZA (Infections and infestations) | 2 (2)
LOCALISED INFECTION (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 11 (11)
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 2 (2)
SEPSIS (Infections and infestations) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 7 (7)
UROSEPSIS (Infections and infestations) | 2 (2)
VIRAL PHARYNGITIS (Infections and infestations) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1)
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1)
EXCORIATION (Injury, poisoning and procedural complications) | 1 (1)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (2)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 2 (2)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 (1)
WOUND (Injury, poisoning and procedural complications) | 1 (1)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1)
HAEMATOCRIT DECREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1)
PROPOFOL INFUSION SYNDROME (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 (1)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1)
NON-HODGKIN'S LYMPHOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MALIGNANT NEOPLASM OF RENAL PELVIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NASAL NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NON-SMALL CELL LUNG CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECURRENT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 (3)
DIZZINESS (Nervous system disorders) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 1 (1)
NEUROTOXICITY (Nervous system disorders) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 3 (3)
PETIT MAL EPILEPSY (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 2 (2)
CONFUSIONAL STATE (Nervous system disorders) | 1 (1)
DEPRESSION (Nervous system disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 4 (5)
URINARY RETENTION (Renal and urinary disorders) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 (4)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 5 (7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PHARYNGEAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PULMONARY OEDEMA (Reproductive system and breast disorders) | 1 (1)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ABDOMINAL HERNIA REPAIR (Surgical and medical procedures) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1)
ANEURYSM (Vascular disorders) | 2 (2)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 3 (3)
AORTIC THROMBOSIS (Vascular disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 2 (2)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 3 (3)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 (2)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 2 (2)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 2 (2)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1)
THROMBOSIS (Vascular disorders) | 2 (2)
VASCULAR STENOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Repair (N=139)
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 (7)
FATIGUE (General disorders) | 9 (9)
PYREXIA (General disorders) | 7 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 (9)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (8)
HAEMATOMA (Vascular disorders) | 8 (10)
HYPOTENSION (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT02393716/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT02393716/SAP_001.pdf